Study Title: Testing whether selected blog posts can improve well-being

Researcher: David Mou MD, Peter Franz, MA

Faculty Advisor: Matt Nock, PhD

Version Date: 11/20/2020

#### **Key Information**

# Why am I being invited to take part in a research study?

We invite you to take part in a research study because we would like to better understand how the articles on TheMighty.com may affect you, especially around the topic of self-harm and suicidal thinking.

#### What should I know about a research study?

- •Whether or not you take part is up to you.
- •Your participation is completely voluntary.
- •You can choose not to take part.
- •You can agree to take part and later change your mind.
- •Your decision will not be held against you.
- •Your refusal to participate will not result in any consequences or any loss of benefits that you are otherwise entitled to receive.
- •You can ask all the questions you want before you decide.

#### Why is this research being done?

Little is known about whether reading materials about suicide affects how people think about suicide. We'd like to understand both how thinking about suicide changes with time, as well as how reading certain articles may affect suicidal thinking.

# How long will the research last and what will I need to do?

We expect that you will be in this research study for two weeks. You will either be sent a daily email with a link to a survey, or you will be sent a link to surveys and articles. Each link will give you detailed instructions.

To the best of your ability, please fill out these surveys the same day you receive them.

Please complete as many of these surveys as possible.

#### Is there any way being in this study could be bad for me?

Very little is known about how reading user-generated articles can affect mood. For some, reading about materials and being asked questions about suicidal ideation may cause emotional distress. You have the right to discontinue the study at any time.

Also, like all websites, there is a risk that your data may be compromised should there be mismanagement of your data.

More detailed information about the study procedures can be found under "What can I expect if I take part in this research."

# Will being in this study help me in any way?

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits include becoming more attentive to how reading certain types of articles affect your mood and the way you think about self-harm. For some, participating may decrease their level of suicidal thinking. This research may also benefit others in that it can help scientists and clinicians better understand what types of articles affect suicidal thinking.

# **Detailed Information**

The following is more detailed information about this study in addition to the information listed above.

# What is the purpose of this research?

Millions of people read articles written by other patients about suicide online. However, little is known whether reading these articles decrease, increase, or have no effect on suicidality. We hope to better understand the effects of reading articles on suicide thinking, with the hope of developing a curriculum of articles that will decrease suicidal thinking in people who read them.

# How long will I take part in this research?

The length of the study will last between 6-8 weeks. A round of the study consists of us sending you a link to your email for 5-14 days, followed by one follow up questionnaire two weeks later. In those we ask you to click on the link and follow the instructions every day. For any given day, the length of activities will be less than 10 minutes. You may be asked to participate in a second round of the study.

#### What can I expect if I take part in this research?

If you agree to participate, we are requesting for your permission to link your data on TheMighty with your data collected as part of this research project. You will be sent an email once a day in the morning, which will include a link that will be specific to you. We ask that you click on the link and fill out the survey. This survey is tailored to you, so please do not forward to anyone else. Sometimes, the surveys may be accompanied by an article on TheMighty.com. These articles focus on the topic of suicide and self-harm. Sometimes, there won't be any accompanying articles.

If you complete at least 75% of the daily surveys, you will be entered into a raffle to receive check for \$250. At the end of the study, we will randomly select two winners to receive these checks. Each daily survey you complete will give you one entry into the raffle, and so the more daily surveys you complete, the greater your chances of winning the raffle.

If you are selected as a winner of the raffle, we will email you to ask for your physical address so we can mail the check. If you cannot provide a physical address, you will not be eligible to win the raffle.

# What happens if I say yes, but I change my mind later?

You can leave the research at any time it will not be held against you. If you choose to withdraw, we will delete your data in order to preserve your privacy.

Is there any way being in this study could be bad for me? (Detailed Risks)

There are some risks you might experience from being in this study. Though there is no scientific evidence, there is a theoretical possibility that reading articles about suicide and/or answering questions about suicidal thinking may increase your suicidal thinking. At any point if you feel uncomfortable, you have the option to quit the study. At the end of each survey, we provide you with information for a suicide hotline.

# If I take part in this research, how will my privacy be protected? What happens to the information you collect?

Efforts will be made to limit the use and disclosure of your Personal Information, including research study records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization. Only TheMighty.com and Harvard University will have access to your data. If identifiers are removed from your identifiable private information that are collected during this research, that information could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

# ClinicalTrials.gov

A description of this research study will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Compensation - If you agree to take part in this research study and complete at least 75% of the daily surveys, you will be entered into a raffle to win a \$250 check. You will be given one entry into the raffle for each day you complete a survey, so the more surveys you complete, the greater your chances of winning. We will notify by email after the data collection is complete to let you know you have won. At that point, we will need you to provide a physical mailing address so we can send you the check. If you cannot provide a physical mailing address, you will not be eligible to win the raffle.

# Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at pfranz@g.harvard.edu.

This research has been reviewed and approved by the Harvard University Area Institutional Review Board ("IRB"). You may talk to them at (617) 496-2847 or cuhs@harvard.edu if:

- •Your questions, concerns, or complaints are not being answered by the research team.
- •You cannot reach the research team.
- •You want to talk to someone besides the research team.
- •You have questions about your rights as a research subject.
- •You want to get information or provide input about this research.